CLINICAL TRIAL: NCT03704064
Title: A Randomized Controlled Trial of Behavioral Weight Loss and Stigma Reduction for Long-Term Weight Loss
Brief Title: Behavioral Weight Loss and Stigma Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rebecca L. Pearl, Ph.D., Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 828274, 202002728; K23HL140176 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: Weight Loss; Weight Stigma; Physical Activity; Cardiovascular Risk Factor
MeSH Terms: conditions — Obesity; Weight Loss; Weight Prejudice; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stigma + BWL Intervention (Experimental): Participants in this group will receive the standard behavioral weight loss (BWL) program, which will be combined with a stigma-reduction intervention (more details provided in the Intervention section). All group meetings will be 90 minutes. Beginning at week 5, the 60-minute BWL sessions will be followed by 30 minutes devoted to stigma-related content. In the monthly and every-other-month weight loss maintenance sessions from weeks 21-72, strategies for coping with weight stigma and challenging internalized beliefs will be reviewed, and participants will be encouraged to use these strategies specifically with physical activity.
  Interventions: Behavioral: Stigma-Reduction Intervention; Behavioral: Behavioral Weight Loss (BWL)
- Standard BWL Intervention (Active Comparator): Participants in this group will be provided with 20 weekly behavioral weight loss (BWL) session (described in more detail in the Intervention section), followed by 6 monthly weight loss maintenance sessions and 3 every-other-month sessions (for a total of 29 visits over 72 weeks). All group meetings will be 90 minutes. Beginning at week 5, BWL content in these sessions will last 60 minutes, with an additional 30 minutes devoted to discussing recipes and food preparation.
  Interventions: Behavioral: Behavioral Weight Loss (BWL)

INTERVENTIONS:
Behavioral: Stigma-Reduction Intervention — Session topics will be based on those tested in a previous pilot study, including: psychoeducation about weight and weight stigma; challenging myths and cognitive distortions related to weight; strategies for coping with instances of stigma; and increasing empowerment and body esteem. The effects of weight stigma on health behaviors will be discussed, and sessions will focus specifically on helping participants overcome stigma-related barriers to physical activity. For example, they will be given strategies to cope with anticipated stigma while exercising in public spaces (e.g., while walking), as well as to challenge self-critical beliefs (e.g., that they are lazy) which may otherwise lead them to avoid exercising. These concrete strategies, along with reducing WBI and improving self-confidence, are intended to increase participants' self-efficacy for and engagement in physical activity.
  Arms: Stigma + BWL Intervention
Behavioral: Behavioral Weight Loss (BWL) — This intervention will be based on the Diabetes Prevention Program. A diet of 1200-1499 calories per day will be prescribed for participants < 250 lb, and 1500-1800 for those ≥ 250 lb. Participants will be instructed to eat a balanced deficit diet. Session topics during the first 20 weeks will include self-monitoring, stimulus control, social support, portion sizes, and goal-setting. Those during weeks 21-72 will focus on skills required for weight loss maintenance and relapse prevention. Physical activity will be begin with a prescription of 60 min/wk, and will gradually progress by 10 minutes over 2-4 week intervals until achieving 150 min/wk by week 20, 200 min/wk by week 46, and 250 min/wk by week 72. Participants will be instructed to spread the activity equally across at least 5 days in bouts that are >10 minutes in duration. Moderate intensity will be prescribed with an emphasis on walking; the vast majority of our research participants self-select this form of activity.

SUMMARY:
This is a randomized controlled trial to test the effects on long-term weight loss of a novel stigma-reduction intervention combined with standard BWL treatment, as compared to BWL alone. Participants will be a total of 104 men and women seeking weight loss, ages 18 years and older, with a body mass index (BMI) of 30 kg/m2 or above (or 27 kg/m2 or above with an obesity-related comorbidity), a history of experiencing weight bias, and elevated levels of WBI. Participants will attend a screening visit in which they will complete a behavioral evaluation with a psychologist and a medical history that will be reviewed by a nurse practitioner or physician. Questionnaires assessing experiences and internalization of weight bias, with confirmation by interviewer assessment during the behavioral evaluation, will be used to determine whether participants meet criteria for having high levels of WBI. Eligible consenting participants will be randomly assigned to the standard BWL intervention (n = 52) or the stigma + BWL intervention (n = 52). All participants will attend weekly, 90-minute group meetings for 20 weeks (20 visits). In the stigma + BWL treatment group, 60 minutes will be devoted to BWL and 30 minutes to weight stigma. In the standard BWL treatment group, the additional 30 minutes will be devoted to sharing recipes and food preparation tips. Following 20 weeks of weight loss treatment, participants will attend group meetings focused on weight loss maintenance, monthly from weeks 21-46 (6 visits), and every-other-month from weeks 47-72 (3 visits). Maintenance sessions in the stigma + BWL group will continue to incorporate discussion of WBI and stigma-related barriers to physical activity. Assessments - which include questionnaires, blood draws, and measurements of body weight and physical activity - will occur at baseline and weeks 20, 46 (no blood draw this week), and 72. Weight will be measured at every group meeting for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be men and women ages 18 years and older.
* Participants must have obesity, defined as a BMI ≥ 30 kg/m2 or ≥ 27 kg/m2 with an obesity-related comorbidity.

  o Obesity-related comorbidities (which confer added CVD risk) will include:
* coronary heart disease;
* other atherosclerotic disease;
* sleep apnea;
* hypercholesteremia (i.e., high cholesterol, as diagnosed by doctor and/or if taking medication to lower cholesterol);
* and components of the metabolic syndrome, including hypertension (SBP ≥130, DBP ≥80 mm Hg, diagnosed by doctor and/or if taking anti-hypertensive medication); fasting blood glucose of 100-125 mg/dL (or prediabetes, diagnosed by doctor),; low HDL cholesterol (<40 mg/dL in men, <50 mg/dL in women), elevated triglycerides (>150 mg/dL, i.e., dyslipidemia diagnosed by doctor or taking medication to treat dyslipidemia), or elevated waist circumference (≥40 in for men, ≥35 in for women),.
* Eligible participants must also report a history of experiencing weight bias as assessed by self-report questionnaire and in-person interview, and have elevated levels of WBI as indicated by an average score of 4 (midpoint) or above on the Weight Bias Internalization Scale (WBIS) and by in-person interview.
* Participants must be seeking weight loss.
* If currently taking medications, dosages must be stable for at least 3 months.
* Participants will be eligible to participate if they exhibit mild to moderate severity of depression, anxiety, or binge eating disorder, as determined by the behavioral evaluation and the screening measures (Beck Depression Inventory-II and Questionnaire for Eating and Weight Patterns; see below for details). Elevated WBIS scores are often associated with these variables.
* Participants taking anti-depressant medication will be eligible if their dose has been stable for a minimum of 3 months.

Eligible female patients will be:

* non-pregnant and non-lactating
* surgically sterile or postmenopausal, or they will agree to continue to use a method of birth control during the study

Participants must:

* have a PCP who is responsible for providing routine care
* have reliable telephone service and/or email access with which to be in contact with the study team
* understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent

Exclusion Criteria:

Applicants will be excluded if they have:

* a diagnosis of type I or II diabetes (for type II diabetes, blood glucose ≥126 mg/dL or A1C ≥6.5);
* uncontrolled hypertension (blood pressure ≥ 160/100 mm Hg);
* experienced a cardiovascular event (e.g., stroke, myocardial infarction) in the last 12 months;
* lost and maintained ≥ 5% of their initial weight in the last 3 months or ≥ 10% in the past 2 years;
* or have participated in individual or group psychotherapy related to weight in the last 3 months (due to the potentially confounding effects of receiving a simultaneous cognitive-behavioral intervention).

  o Participants who have recently received or are currently receiving therapy for a pre-existing mental health issue unrelated to weight (e.g., psychotherapy for depression or anxiety, or marriage, grief, or career counseling) may be eligible if the therapy is deemed by the Principal Investigator to be unlikely to affect weight, eating habits, or physical activity.
* Applicants with severe symptoms of mood (BDI-II score ≥ 29), anxiety, or binge eating disorder, and any severity of thought or substance use disorders will not be accepted into the study, as these symptoms may interfere with individuals' ability to adhere to a weight loss program.

  o Clinician judgment will be used to determine severity of mood disorder symptoms independent from obesity-related concerns and complications (e.g., fatigue), and decisions about applicants' eligibility based on psychiatric symptoms will fall within the Principal Investigator's discretion.
* Individuals with bulimia nervosa will not be eligible to participate, because weight loss may be contraindicated.
* Applicants with current, active suicidal ideation, and/or a suicide attempt within the past year will be excluded from the study and referred to psychiatric treatment facilities in the greater Philadelphia area.
* Applicants will not be eligible if they have a history of bariatric surgery.
* Women who are nursing, pregnant, or planning to become pregnant in the next 16 months are not eligible to participate.
* Applicants who report obtaining 150 minutes or more of structured physical activity per week (e.g., 30 minutes 5 days per week) will not be eligible, as they will already be obtaining the recommended amount of physical activity and may not be able to further increase their activity as part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Pearl, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- The University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Sheynblyum M, Wadden TA, Latner JD, Pearl RL. Longitudinal associations of internalized weight stigma with physical activity and weight loss. Obes Sci Pract. 2024 Jul 3;10(4):e773. doi: 10.1002/osp4.773. eCollection 2024 Aug. PMID 38966255
- [Derived] Pearl RL, Wadden TA, Bach C, LaFata EM, Gautam S, Leonard S, Berkowitz RI, Latner JD, Jakicic JM. Long-term effects of an internalized weight stigma intervention: A randomized controlled trial. J Consult Clin Psychol. 2023 Jul;91(7):398-410. doi: 10.1037/ccp0000819. Epub 2023 May 8. PMID 37155264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Started | 52 | 53
Week 20 | 44 | 46
Week 46 | 44 | 46
Week 72 | 42 | 47
Completed | 42 | 47
Not Completed | 10 | 6
Not completed — Lost to Follow-up | 8 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — No longer available for study visits | 0 | 1
Not completed — Censoring event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.96 (12.86) | 49.15 (12.05) | 49.06 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 46 | 95
  Male | 3 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 52 | 50 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 37 | 37 | 74
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 104.39 (18.21) | 104.48 (21.04) | 104.44 (19.59)
Height [Mean (Standard Deviation); unit: cm] | 165.04 (7.13) | 166.35 (7.87) | 165.70 (7.51)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 38.23 (5.59) | 37.48 (5.16) | 37.85 (5.36)

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change at Week 72
Description: Estimated mean percent change in weight from baseline to week 72
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: percent weight change
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
percent weight change | -7.16 (0.95) | -5.19 (0.92)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Net) = -1.97, Standard Error of Mean 1.32

2. Secondary Outcome: Loss of 5% or Greater of Initial Body Weight at Week 72
Description: The percentage of participants who lost 5% or greater of their initial body weight at week 72
Time Frame: Baseline to week 72
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 20 | 21
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.89, Mixed Models Analysis; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.4 to 3.4]

3. Secondary Outcome: Loss of 10% or Greater of Initial Body Weight at Week 72
Description: The percentage of participants who lost 10% or greater of their initial body weight at week 72
Time Frame: Baseline to week 72
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 14 | 7
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.06, Mixed Models Analysis; Odds Ratio (OR) = 3.7, 95% CI 2-sided [1.0 to 14.7]

4. Secondary Outcome: Percent Weight Change at Week 46
Description: Estimated mean percent weight change
Time Frame: Baseline to week 46
Measure: Mean (Standard Error); unit: percent weight change
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
percent weight change | -8.2 (0.9) | -5.9 (0.9)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = -2.4, Standard Error of Mean 1.3

5. Secondary Outcome: Percent Weight Change at Week 20
Description: Estimated mean percent weight change
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: percent weight change
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
percent weight change | -6.7 (0.9) | -5.7 (0.9)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.42, Mixed Models Analysis; Mean Difference (Net) = -1.1, Standard Error of Mean 1.3

6. Secondary Outcome: Loss of 5% or Greater of Initial Body Weight at Week 46
Description: The percentage of participants who lost 5% or greater of their initial body weight at week 46
Time Frame: Baseline to week 46
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 28 | 22
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.24, Mixed Models Analysis; Odds Ratio (OR) = 2.0, 95% CI 2-sided [0.6 to 6.3]

7. Secondary Outcome: Loss of 10% or Greater of Initial Body Weight at Week 46
Description: The percentage of participants who lost 10% or greater of their initial body weight at week 46
Time Frame: Baseline to week 46
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 15 | 9
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.24, Mixed Models Analysis; Odds Ratio (OR) = 2.2, 95% CI 2-sided [0.6 to 8.1]

8. Secondary Outcome: Loss of 5% or Greater of Initial Body Weight at Week 20
Description: The percentage of participants who lost 5% or greater of their initial body weight at week 20
Time Frame: Baseline to week 20
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 31 | 22
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.07, Mixed Models Analysis; Odds Ratio (OR) = 3.0, 95% CI 2-sided [0.9 to 9.6]

9. Secondary Outcome: Loss of 10% or Greater of Initial Body Weight at Week 20
Description: The percentage of participants who lost 10% or greater of their initial body weight at week 20
Time Frame: Baseline to week 20
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 11 | 5
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.21, Mixed Models Analysis; Odds Ratio (OR) = 2.6, 95% CI 2-sided [0.6 to 11.4]

10. Secondary Outcome: Change in Minutes of Physical Activity (Accelerometer) at Week 72
Description: Estimated mean change in daily minutes of physical activity, as measured by accelerometry
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: Minutes per day
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Minutes per day
  MVPA per day with 10 minute bouts | 9.6 (4.1) | 7.2 (4.1)
  MVPA per day with 20 minute bouts | 9.4 (3.2) | 8.4 (3.1)
  Moderate activity per day | 3.2 (6.8) | -10.2 (6.7)
  Light activity per day | -35.6 (15.1) | -51.5 (14.3)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; MVPA per day with 10 minute bouts; Test type: Superiority; p = 0.62, Mixed Models Analysis; Mean Difference (Net) = 2.4, Standard Error of Mean 5.8
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; MVPA per day with 20 minute bouts; Test type: Superiority; p = 0.92, Mixed Models Analysis; Mean Difference (Net) = 1.0, Standard Error of Mean 4.5
Statistical Analysis 3: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Moderate activity per day; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = 13.4, Standard Error of Mean 9.6
Statistical Analysis 4: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Light activity per day; Test type: Superiority; p = 0.41, Mixed Models Analysis; Mean Difference (Net) = 15.9, Standard Error of Mean 20.8

11. Secondary Outcome: Change in Minutes of Physical Activity (Accelerometer) at Week 46
Description: Estimated mean change in daily minutes of physical activity, as measured by accelerometry
Time Frame: Baseline to week 46
Measure: Mean (Standard Error); unit: Minutes per day
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Minutes per day
  MVPA per day with 10 minute bouts | 9.5 (4.3) | 5.4 (4.4)
  MVPA per day with 20 minute bouts | 9.9 (3.4) | 10.5 (3.2)
  Moderate activity per day | 0.6 (7.2) | -17.9 (7.2)
  Light activity per day | -37.1 (15.9) | -67.0 (16.0)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; MVPA per day with 10 minute bouts; Test type: Superiority; p = 0.46, Mixed Models Analysis; Mean Difference (Net) = 4.1, Standard Error of Mean 6.1
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; MVPA per day with 20 minute bouts; Test type: Superiority; p = 0.87, Mixed Models Analysis; Mean Difference (Net) = -0.5, Standard Error of Mean 4.9
Statistical Analysis 3: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Moderate activity per day; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = 18.5, Standard Error of Mean 10.1
Statistical Analysis 4: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Light activity per day; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Net) = 30.0, Standard Error of Mean 22.5

12. Secondary Outcome: Change in Minutes of Physical Activity (Accelerometer) at Week 20
Description: Estimated mean change in daily minutes of physical activity, as measured by accelerometry
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: Minutes per day
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Minutes per day
  MVPA per day with 10 minute bouts | 11.4 (4.0) | 8.8 (4.1)
  MVPA per day with 20 minute bouts | 10.5 (2.6) | 9.9 (2.7)
  Moderate activity per day | 10.6 (6.7) | 4.7 (6.7)
  Light activity per day | -19.0 (14.2) | 3.8 (13.2)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; MVPA per day with 10 minute bouts; Test type: Superiority; p = 0.63, Mixed Models Analysis; Mean Difference (Net) = 2.2, Standard Error of Mean 5.7
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; MVPA per day with 20 minute bouts; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Net) = 0.6, Standard Error of Mean 3.7
Statistical Analysis 3: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Moderate activity per day; Test type: Superiority; p = 0.52, Mixed Models Analysis; Mean Difference (Net) = 6.0, Standard Error of Mean 9.4
Statistical Analysis 4: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Light activity per day; Test type: Superiority; p = 0.27, Mixed Models Analysis; Mean Difference (Net) = -21.8, Standard Error of Mean 19.4

13. Secondary Outcome: Change in Energy Expenditure at Week 72
Description: Estimated mean change in energy expenditure, as measured by the Paffenbarger Physical Activity Questionnaire. Higher kilocalories (kcal) indicate greater energy expenditure.
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: Kcal
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Kcal | 314.8 (105.9) | 307.5 (108.0)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.84, Mixed Models Analysis; Mean Difference (Net) = 7.3, Standard Error of Mean 151.2

14. Secondary Outcome: Change in Energy Expenditure at Week 46
Description: as for outcome 13
Time Frame: Baseline to week 46
Measure: Mean (Standard Error); unit: Kcal
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Kcal | 148.7 (90.1) | 260.4 (103.5)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.53, Mixed Models Analysis; Mean Difference (Net) = -111.7, Standard Error of Mean 137.2

15. Secondary Outcome: Change in Energy Expenditure at Week 20
Description: as for outcome 13
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: Kcal
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Kcal | 452.5 (111.9) | 289.3 (105.6)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.27, Mixed Models Analysis; Mean Difference (Net) = 163.2, Standard Error of Mean 154.0

16. Secondary Outcome: Change in Exercise Self-efficacy at Week 72
Description: Estimated mean change on the Self-Efficacy to Exercise Scale (total score 0-90; higher scores = greater self-efficacy)
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | -9.4 (3.3) | -15.0 (3.2)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.22, Mixed Models Analysis; Mean Difference (Net) = 5.7, Standard Error of Mean 4.6

17. Secondary Outcome: Change in Exercise Self-efficacy at Week 46
Description: Estimated mean change on the Self-Efficacy to Exercise Scale (total score 0-90; higher scores = greater self-efficacy)
Time Frame: Baseline to week 46
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | -10.6 (3.2) | -15.9 (3.2)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.24, Mixed Models Analysis; Mean Difference (Net) = 5.3, Standard Error of Mean 4.6

18. Secondary Outcome: Change in Exercise Self-efficacy at Week 20
Description: Estimated mean change on the Self-Efficacy to Exercise Scale (total score 0-90; higher scores = greater self-efficacy)
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | 1.1 (3.2) | -2.0 (3.1)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = 3.2, Standard Error of Mean 4.5

19. Secondary Outcome: Change in Eating Self-efficacy at Week 72
Description: Estimated mean change on the Weight Efficacy Lifestyle Questionnaire - Short Form (total score 0-72; higher scores = greater self-efficacy)
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | 6.5 (2.5) | 1.7 (2.4)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = 4.9, Standard Error of Mean 3.4

20. Secondary Outcome: Change in Eating Self-efficacy at Week 46
Description: as for outcome 19
Time Frame: Baseline to week 46
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | 5.8 (2.4) | -1.0 (2.4)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.045, Mixed Models Analysis; Mean Difference (Net) = 6.8, Standard Error of Mean 3.4

21. Secondary Outcome: Change in Eating Self-efficacy at Week 20
Description: as for outcome 19
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | 12.3 (2.4) | 8.6 (2.3)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.27, Mixed Models Analysis; Mean Difference (Net) = 3.7, Standard Error of Mean 3.4

22. Secondary Outcome: Change in Triglycerides at Week 72
Description: Estimated mean change in triglyceride concentration in blood
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
mg/dL | -9.9 (6.4) | -13.7 (6.8)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Net) = 3.9, Standard Error of Mean 9.4

23. Secondary Outcome: Change in Triglycerides at Week 20
Description: Estimated mean change in triglyceride concentration in blood
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
mg/dL | -10.9 (6.3) | -7.7 (6.5)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.67, Mixed Models Analysis; Mean Difference (Net) = -3.3, Standard Error of Mean 9.1

24. Secondary Outcome: Change in Blood Pressure at Week 72
Description: Estimated mean change in blood pressure (systolic blood pressure and diastolic blood pressure; mmHg)
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
mmHg
  Systolic Blood Pressure | -5.0 (1.7) | -5.6 (1.8)
  Diastolic Blood Pressure | -1.9 (1.1) | -2.0 (1.1)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Systolic Blood Pressure; Test type: Superiority; p = 0.80, Mixed Models Analysis; Mean Difference (Net) = 0.6, Standard Error of Mean 2.5
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Diastolic Blood Pressure; Test type: Superiority; p = 0.94, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 1.1

25. Secondary Outcome: Change in Blood Pressure Week 20
Description: Estimated mean change in blood pressure (systolic blood pressure and diastolic blood pressure; mmHg)
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: mmHG
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
mmHG
  Systolic Blood Pressure | -9.7 (1.7) | -5.4 (1.6)
  Diastolic Blood Pressure | -3.5 (1.1) | -3.6 (1.1)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Systolic Blood Pressure; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = -4.3, Standard Error of Mean 2.3
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Diastolic Blood Pressure; Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 1.5

26. Secondary Outcome: Change in Weight Bias Internalization Scale Score at Week 72
Description: Estimated mean change score on the Weight Bias Internalization Scale (scale scoring 1-7; higher scores indicate greater weight bias internalization).
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | -1.7 (0.2) | -1.5 (0.1)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.30, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.2

27. Secondary Outcome: Change in Weight Bias Internalization Scale Score at Week 46
Description: as for outcome 26
Time Frame: Baseline to week 46
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | -1.5 (0.1) | -1.4 (0.1)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.67, Mixed Models Analysis; Mean Difference (Net) = -0.1, Standard Error of Mean 0.2

28. Secondary Outcome: Change in Weight Bias Internalization Scale Score at Week 20
Description: as for outcome 26
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale | -1.4 (0.1) | -1.2 (0.1)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.45, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.2

29. Secondary Outcome: "Remission" of Elevated Weight Bias Internalization at Week 72
Description: Percentage of participants who score below 4.0 on the Weight Bias Internalization Scale (scale scoring 1-7; higher scores indicate greater weight bias internalization)
Time Frame: Baseline to week 72
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 28 | 26
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.38, Mixed Models Analysis; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.5 to 5.9]

30. Secondary Outcome: "Remission" of Elevated Weight Bias Internalization at Week 46
Description: as for outcome 29
Time Frame: Baseline to week 46
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 24 | 25
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.95, Mixed Models Analysis; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.3 to 3.3]

31. Secondary Outcome: "Remission" of Elevated Weight Bias Internalization at Week 20
Description: as for outcome 29
Time Frame: Baseline to week 20
Measure: Count of Participants; unit: Participants
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
Participants | 25 | 26
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Test type: Superiority; p = 0.99, Mixed Models Analysis; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.3 to 3.1]

32. Secondary Outcome: Change in Weight Self-stigma Scores at Week 72
Description: Estimated mean change score for Total score (WSSQ-Total, summed 12-60) and two subscales of Self-Devaluation (WSSQ-SD) and Fear of Enacted Stigma (WSSQ-FE) (summed 6-30); higher scores indicate greater weight self-stigma.
Time Frame: Baseline to week 72
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale
  WSSQ-Total | -9.7 (1.1) | -6.7 (1.1)
  WSSQ-SD | -5.0 (0.7) | -3.8 (0.6)
  WSSQ-FE | -4.7 (0.7) | -2.9 (0.7)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-Total; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Net) = -3.0, Standard Error of Mean 1.6
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-SD; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Net) = -1.8, Standard Error of Mean 0.9
Statistical Analysis 3: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-FE; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Net) = -1.2, Standard Error of Mean 0.9

33. Secondary Outcome: Change in Weight Self-stigma Scores at Week 46
Description: as for outcome 32
Time Frame: Baseline to week 46
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale
  WSSQ-Total | -8.5 (1.1) | -5.5 (1.1)
  WSSQ-SD | -4.0 (0.7) | -2.8 (0.6)
  WSSQ-FE | -4.5 (0.6) | -2.7 (0.6)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-Total; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Net) = -3.0, Standard Error of Mean 1.5
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-SD; Test type: Superiority; p = 0.18, Mixed Models Analysis; Mean Difference (Net) = -1.2, Standard Error of Mean 0.9
Statistical Analysis 3: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-FE; Test type: Superiority; p = 0.046, Mixed Models Analysis; Mean Difference (Net) = -1.8, Standard Error of Mean 0.9

34. Secondary Outcome: Change in Weight Self-stigma Scores at Week 20
Description: as for outcome 32
Time Frame: Baseline to week 20
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 52 | 53
score on a scale
  WSSQ-Total | -8.2 (1.1) | -5.5 (1.1)
  WSSQ-SD | -4.6 (0.7) | -3.2 (0.6)
  WSSQ-FE | -3.6 (0.6) | -2.3 (0.6)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-Total; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = -2.7, Standard Error of Mean 1.5
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-SD; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Net) = -1.5, Standard Error of Mean 0.9
Statistical Analysis 3: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; WSSQ-FE; Test type: Superiority; p = 0.15, Mixed Models Analysis; Mean Difference (Net) = -1.3, Standard Error of Mean 0.9

35. Secondary Outcome: Treatment Acceptability at Week 20
Description: To assess treatment acceptability, participants in both groups rated (1-7) how acceptable and helpful the program was, how much they liked the program, and how satisfied they were; scores for these 4 items were averaged. Participants also rated (1-7) the BWL treatment, as well as the stigma intervention (i.e., BIAS component) or recipe exchange, on how helpful they found each component of the program, how much they liked the components, and how much they learned. Scores for these three items were averaged (1-7) separately for the BWL treatment, BIAS component, and recipe exchange. Participants rated how much they learned BWL scores, and how much they learned and used skills related to stigma (all averaged 1-7). Higher scores indicate greater treatment acceptability.
Time Frame: Week 20
Population: Participants randomized to the stigma + BWL group did not receive (and thus did not rate) the recipe exchange component of treatment. Participants in the Standard BWL group did not receive (and did not rate) the BIAS treatment component.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 44 | 48
score on a scale
  Overall treatment acceptability | 6.4 (0.2) | 5.8 (0.2)
  BWL component acceptability | 6.1 (0.2) | 5.9 (0.2)
  BIAS vs recipe component acceptability | 6.1 (0.2) | 4.6 (0.2)
  BWL skill acquisition | 6.2 (0.2) | 5.6 (0.2)
  Stigma-related skill acquisition | 5.8 (0.2) | 4.9 (0.2)
  Stigma-related skill use | 4.1 (0.1) | 3.3 (0.1)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Overall treatment acceptability; Test type: Superiority; p = 0.04, ANOVA; Mean Difference (Net) = 0.6, Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; BWL component acceptability; Test type: Superiority; p = 0.35, ANOVA; Mean Difference (Net) = 0.3, Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; BIAS vs recipe component acceptability; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Net) = 1.5, Standard Error of Mean 0.3
Statistical Analysis 4: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; BWL skill acquisition; Test type: Superiority; p = 0.01, ANOVA; Mean Difference (Net) = 0.6, Standard Error of Mean 0.2
Statistical Analysis 5: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Stigma-related skill acquisition; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Net) = 1.0, Standard Error of Mean 0.3
Statistical Analysis 6: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Stigma-related skill use; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Net) = 0.7, Standard Error of Mean 0.2

36. Secondary Outcome: Treatment Acceptability at Week 72
Description: as for outcome 35
Time Frame: Week 72
Population: as for outcome 35
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
Number analyzed (Participants) | 41 | 44
score on a scale
  Overall treatment acceptability | 6.1 (0.2) | 5.8 (0.2)
  BWL component acceptability | 6.0 (0.2) | 5.7 (0.2)
  BIAS vs recipe component acceptability | 5.9 (0.3) | 4.1 (0.3)
  BWL skill acquisition | 5.9 (0.2) | 5.6 (0.2)
  Stigma-related skill acquisition | 5.8 (0.2) | 5.0 (0.2)
  Stigma-related skill use | 3.8 (0.1) | 3.3 (0.1)
Statistical Analysis 1: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Overall treatment acceptability; Test type: Superiority; p = 0.24, ANOVA; Mean Difference (Net) = 0.3, Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; BWL component acceptability; Test type: Superiority; p = 0.28, ANOVA; Mean Difference (Net) = 0.3, Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; BIAS vs recipe component acceptability; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Net) = 1.8, Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; BWL skill acquisition; Test type: Superiority; p = 0.34, ANOVA; Mean Difference (Net) = 0.3, Standard Error of Mean 0.3
Statistical Analysis 5: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Stigma-related skill acquisition; Test type: Superiority; p = 0.008, ANOVA; Mean Difference (Net) = 0.8, Standard Error of Mean 0.3
Statistical Analysis 6: Comparison: Stigma + BWL Intervention vs Standard BWL Intervention; Stigma-related skill use; Test type: Superiority; p = 0.001, ANOVA; Mean Difference (Net) = 0.6, Standard Error of Mean 0.2

37. Other Pre Specified Outcome: Change in Minutes of Sedentary Time at Week 72
Description: Single item from Global Physical Activity Questionnaire (minutes)
Time Frame: Baseline to week 72
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Change in Minutes of Sedentary Time at Week 46
Description: Single item from Global Physical Activity Questionnaire (minutes)
Time Frame: Baseline to week 46
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Change in Minutes of Sedentary Time at Week 20
Description: Single item from Global Physical Activity Questionnaire (minutes)
Time Frame: Baseline to week 20
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Change in High-density Lipoprotein (HDL) Cholesterol at Week 72
Description: Concentration in blood, controlling for medication use
Time Frame: Baseline to week 72
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Change in High-density Lipoprotein (HDL) Cholesterol at Week 20
Description: Concentration in blood, controlling for medication use
Time Frame: Baseline to week 20
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Change in Waist Circumference at Week 72
Time Frame: Baseline to week 72
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Change in Waist Circumference at Week 20
Time Frame: Baseline to week 20
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Change in Blood Glucose at Week 72
Description: Concentration in blood, controlling for medication use
Time Frame: Baseline to week 72
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Change in Blood Glucose at Week 20
Description: Concentration in blood, controlling for medication use
Time Frame: Baseline to week 20
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Change in C-reactive Protein at Week 72
Description: Concentration in blood
Time Frame: Baseline to week 72
Reporting Status: Not Posted

47. Other Pre Specified Outcome: Change in C-reactive Protein at Week 20
Description: Concentration in blood
Time Frame: Baseline to week 20
Reporting Status: Not Posted

48. Other Pre Specified Outcome: Change in Stereotype Endorsement Scores at Week 72
Description: Fat Phobia Scale (scores averaged 1-5, with higher scores indicating greater weight bias)
Time Frame: Baseline to week 72
Reporting Status: Not Posted

49. Other Pre Specified Outcome: Change in Stereotype Endorsement Scores at Week 46
Description: Fat Phobia Scale (scores averaged 1-5, with higher scores indicating greater weight bias)
Time Frame: Baseline to week 46
Reporting Status: Not Posted

50. Other Pre Specified Outcome: Change in Stereotype Endorsement Scores at Week 20
Description: Fat Phobia Scale (scores averaged 1-5, with higher scores indicating greater weight bias)
Time Frame: Baseline to week 20
Reporting Status: Not Posted

51. Other Pre Specified Outcome: Change in Weight-related Quality of Life at Week 72
Description: Impact of Weight on Quality of Life Questionnaire-Lite (total score and 5 subscales; t-scores ranging from 0-100, with higher scores indicating better quality of life)
Time Frame: Baseline to week 72
Reporting Status: Not Posted

52. Other Pre Specified Outcome: Change in Weight-related Quality of Life at Week 46
Description: as for outcome 51
Time Frame: Baseline to week 46
Reporting Status: Not Posted

53. Other Pre Specified Outcome: Change in Weight-related Quality of Life at Week 20
Description: as for outcome 51
Time Frame: Baseline to week 20
Reporting Status: Not Posted

54. Other Pre Specified Outcome: Change in Perceived Stress at Week 72
Description: Perceived Stress Scale (total score 0-40; higher scores = greater perceived stress)
Time Frame: Baseline to week 72
Reporting Status: Not Posted

55. Other Pre Specified Outcome: Change in Perceived Stress at Week 46
Description: Perceived Stress Scale (total score 0-40; higher scores = greater perceived stress)
Time Frame: Baseline to week 46
Reporting Status: Not Posted

56. Other Pre Specified Outcome: Change in Perceived Stress at Week 20
Description: Perceived Stress Scale (total score 0-40; higher scores = greater perceived stress)
Time Frame: Baseline to week 20
Reporting Status: Not Posted

57. Other Pre Specified Outcome: Change in Depression Symptoms at Week 72
Description: Patient Health Questionnaire-9 (scores summed 0-27; higher scores = more symptoms of depression)
Time Frame: Baseline to week 72
Reporting Status: Not Posted

58. Other Pre Specified Outcome: Change in Depression Symptoms at Week 46
Description: Patient Health Questionnaire-9 (scores summed 0-27; higher scores = more symptoms of depression)
Time Frame: Baseline to week 46
Reporting Status: Not Posted

59. Other Pre Specified Outcome: Change in Depression Symptoms at Week 20
Description: Patient Health Questionnaire-9 (scores summed 0-27; higher scores = more symptoms of depression)
Time Frame: Baseline to week 20
Reporting Status: Not Posted

60. Other Pre Specified Outcome: Change in Body Image Scores at Week 72
Description: Body Appreciation Scale (scores averaged 1-5; higher scores = greater body appreciation)
Time Frame: Baseline to week 72
Reporting Status: Not Posted

61. Other Pre Specified Outcome: Change in Body Image Scores at Week 46
Description: Body Appreciation Scale (scores averaged 1-5; higher scores = greater body appreciation)
Time Frame: Baseline to week 46
Reporting Status: Not Posted

62. Other Pre Specified Outcome: Change in Body Image Scores at Week 20
Description: Body Appreciation Scale (scores averaged 1-5; higher scores = greater body appreciation)
Time Frame: Baseline to week 20
Reporting Status: Not Posted

63. Other Pre Specified Outcome: Change in Presence and Frequency of Binge Eating at Week 72
Description: Questionnaire on Eating and Weight Patterns (yes/no and episodes per week)
Time Frame: Baseline to week 72
Reporting Status: Not Posted

64. Other Pre Specified Outcome: Change in Presence and Frequency of Binge Eating at Week 46
Description: Questionnaire on Eating and Weight Patterns (yes/no and episodes per week)
Time Frame: Baseline to week 46
Reporting Status: Not Posted

65. Other Pre Specified Outcome: Change in Presence and Frequency of Binge Eating at Week 20
Description: Questionnaire on Eating and Weight Patterns (yes/no and episodes per week)
Time Frame: Baseline to week 20
Reporting Status: Not Posted

66. Other Pre Specified Outcome: Change in Self-monitoring Behaviors at Week 72
Description: Food records and self-report recording of food intake and physical activity
Time Frame: Baseline to week 72
Reporting Status: Not Posted

67. Other Pre Specified Outcome: Change in Self-monitoring Behaviors at Week 46
Description: Food records and self-report recording of food intake and physical activity
Time Frame: Baseline to week 46
Reporting Status: Not Posted

68. Other Pre Specified Outcome: Change in Self-monitoring Behaviors at Week 20
Description: Food records and self-report recording of food intake and physical activity
Time Frame: Baseline to week 20
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through week 72
Description: At each contact with participants, study personnel non-systematically collected information on any adverse events (AEs) self-reported by participants. In addition, AEs were systematically assessed at the scheduled assessments. AEs were documented by study staff in consultation with a nurse practitioner and/or physician. Serious adverse events (SAEs) were reported immediately to the study sponsor, Data and Safety Monitor, and the Institutional Review Board.
Arm/Group | Stigma + BWL Intervention | Standard BWL Intervention
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 14/52 | 17/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stigma + BWL Intervention (N=52) | Standard BWL Intervention (N=53)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Knee pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Contact dermatitis (Product Issues) | 4 (4) | 2 (2) — Skin irritation on wrist from wearing accelerometer wristband
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
Viral gastroenteritis (Infections and infestations) | 3 (3) | 7 (7)
Migraine (Nervous system disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT03704064/Prot_SAP_006.pdf
  • Informed Consent Form (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03704064/ICF_007.pdf